CLINICAL TRIAL: NCT00896441
Title: Functional MRI Before and After Treatment for Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Clinical Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-04202009-2339; Stanford IRB #15305 (Other: Stanford University Institutional Review Board)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Depression; Mood Disorders; Depressive Disorder
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed patients (Experimental): Depressed patients assigned in an open-label study of citalopram
  Interventions: Drug: Citalopram
- Controls (No Intervention): Healthy controls used as a comparison (no intervention) group for change in resting-state fMRI over time

INTERVENTIONS:
Drug: Citalopram — Refer to Detailed Description Section for full description of intervention. Week 1 (baseline): Subject will complete several tests to assess the subject's memory and concentration. Following visit, they will begin treatment with the antidepressant citalopram.
  Week 1 MRI: Subject will have their first MRI. Week 2 visit: Physician will meet with they to assess the subject's overall condition.
  Week 2 MRI: Subject will have the subject's second MRI. Week 4 visit: The study physician will meet with the subject to assess their overall condition.
  Week 6 (Telephone check-in): The study physician will check in with the subject by telephone to assess the subject's overall condition.
  Week 8: (End-of-study visit) Subject will take repeated tests of memory and concentration. The study physician will also discuss recommendations for further treatment of the subject's depression.
  Week 8 MRI: Around the time of the subject's week 8 visit they will have the subject's third and final MRI.
  Arms: Depressed patients

SUMMARY:
The purpose of this study is to help us understand how depression changes brain activity and how this relates to mood, anxiety, and cognitive functions like memory. We also hope to develop a brain imaging test that will predict either before or within two weeks of starting a medicine whether the treatment will work.

DETAILED DESCRIPTION:
You were selected as a possible participant because you are suffering from a major depressive episode, and you have not previously tried the medication used in this study to treat depression. Approximately 60 subjects will participate in this study: 30 subjects who are currently suffering from a major depressive episode and 30 subjects who have never suffered from a major depressive episode.

If you choose to participate, you will be seen at the clinic for a total of five times plus three MRI scans. You will be seen once for a screening visit. If you choose to enroll, you will return a week later for the baseline visit and again at weeks 2, 4 and 8. Around the time of week one (baseline), week 2 and week 8 you will also undergo an MRI scan of the brain.

Screening Visit: The study physician and the research study staff will first screen you for eligibility. The screening visit includes meeting with a physician for a discussion of your medical history and current medications, taking your blood pressure, and checking your weight. Women of childbearing potential will also have a urine pregnancy test. You will meet with a member of the research staff for an interview to collect information about your depression and other psychiatric symptoms you have experienced. The purpose of the interview is to confirm your diagnosis and assess the current severity of your depression. The screening visit will take approximately 2 hours.

Week 1 (baseline): If you are eligible to continue with the study, you will return to the clinic within 7 days for a baseline visit. At your baseline visit, you will complete several tests to assess your memory and concentration. These tests are being conducted because problems with memory and concentration are common in people who are depressed and the researchers want to find out if there is a difference in your memory and concentration before and after taking the study medication. We also wish to compare the results to any findings from the brain imaging. Following the baseline visit, you will begin treatment with the antidepressant citalopram. The starting dose is 20 mg once per day.

Week 1 MRI: Around the time of your week one (baseline) visit and before starting medications, you will have your first MRI.

Week 2 visit: At the end of your second week, the study physician will meet with you to assess your overall condition. Your antidepressant medication will be counted to verify that you have been taking it as prescribed. Your dose will likely not change, but it is possible that it will be increased to as much as 40 mg. If you are experiencing side effects, your dose may be decreased. We will provide you with enough medication to last until your next visit.

Week 2 MRI: Around the time of your week 2 visit you will have your second MRI.

Week 4 visit: The study physician will meet with you to assess your overall condition. Your antidepressant medication will be counted to verify that you have been taking it as prescribed. The dose may be left unchanged, increased up to a total of 40 mg daily or decreased, if you are experiencing side effects (to a minimum of 20 mg daily). You will also be asked about any other medications you have taken since your last visit. We will provide you with enough medication to last until your next visit.

Week 6 (Telephone check-in): The study physician will check in with you by telephone to assess your overall condition. The dose of the citalopram may be left unchanged, increased to a maximum of 60 mg daily or decreased (to a minimum to 20 m daily) if you are experiencing side effects.

Week 8: (End-of-study visit) In addition to the usual visit procedures, the end-of-study visit will include repeated tests of memory and concentration. The study physician will also discuss recommendations for further treatment of your depression. No study medication will be dispensed at this visit.

Week 8 MRI: Around the time of your week 8 visit you will have your third and final MRI.

ELIGIBILITY:
Inclusion Criteria:

Patients will be aged 18-65, have no significant neurologic history, must meet DSM-IV criteria for a diagnosis of major depression and be free of antidepressant or other psychotropic medication for a minimum of two weeks before enrollment. If a subject is talking psychiatric medication he/she may be weaned off of the medication by their treating physician prior to study enrollment. Such a course of action would only be advised if the current medication was not considered to be of any benefit to the subject. In particular, if a patient is on antidepressant medication which is of benefit, we would not advise tapering off medication -- and subsequent risk of relapse -- in order to participate in the study. The same line of thinking applies to all psychiatric diagnoses and associated medications candidate subjects may be taking.

Exclusion Criteria:

1. Significant head trauma with loss of consciousness.
2. Active abuse of alcohol or illegal substances.
3. Excluded psychiatric diagnoses include: Bipolar Affective Disorder, primary psychotic disorders (Schizophrenia, Schizoaffective disorder), Obsessive-Compulsive Disorder
4. Pregnant or nursing women.
5. Any contraindication to being scanned in the 3T scanner at the Lucas Center such as having a pacemaker or any implanted device that has not been cleared for scanning at 3 Tesla.
6. Any significant neurologic history (i.e. seizure, stroke, multiple sclerosis).
7. Use of psychotropic medications within 2 weeks of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-02; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Greicius, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants in the Healthy controls group withdrew consent prior to allocation to study arm.
Groups:
- Depressed: Depressed individuals
- Healthy Controls: Participants with no history of psychiatric illness
Period: Overall Study
Arm/Group | Depressed | Healthy Controls
Started | 17 | 9
Completed | 15 | 9
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: 2 participants in the Depressed arm who did not complete study per protocol are not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Depressed | Healthy Controls | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.00 (12.6) | 31.92 (11.2) | 36.50 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale Percent Change From Day 0 to D56
Description: Utilized the Hamilton Depression Rating Scale (HAM), 21-item version to assess depressive symptoms, with a range of 0-63. Higher scores indicate more depression. For the change score, it is Baseline less Day 56 HAM total / Baseline. Thus, larger values mean a greater decrease in the level of depression
Time Frame: % change from baseline to Day 56 ( week 8)
Population: Only participants completing the protocol are included in the analysis; thus, the N = 12. Only participants in the Depressed group were analyzed for change in depressive symptoms.
Measure: Mean (Standard Deviation); unit: percentage of change in depression
Arm/Group | Depressed
Number analyzed (Participants) | 12
percentage of change in depression | .4125 (.26)
Statistical Analysis 1: Comparison: Depressed; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; One sample t-test

2. Primary Outcome: Voxel-wise Changes in Resting State Functional Connectivity to the Posterior Cingulate Cortex
Description: The dependent variable, measured in more than 30,000 voxels across the whole brain, was the functional connectivity between the posterior cingulate cortex seed region and each voxel. This is derived as the correlation coefficient between the blood-oxygen-level dependent (BOLD) signal timeseries in the seed region and the BOLD signal timeseries in each voxel.
Time Frame: baseline and week 8
Population: Owing to the limited sample size, we first examined this measure in the depressed subjects using a paired-sample t-test at each of the 30,000+ voxels. No significant voxels were detected in this analysis and so subsequent analyses combining the depressed subjects and the healthy control subjects in a single model were not performed.
Measure: Number; unit: significant voxels
Arm/Group | Depressed
Number analyzed (Participants) | 13
significant voxels | 0

3. Secondary Outcome: Hamilton Anxiety Scale
Description: Hamilton Anxiety Scale (HAMA) was utilized. Scores range from 0-56, with higher scores indicating more anxiety. The change score utilized baseline and Day 56 (week 8) scores. The change scores was HAMA day 1 less Ham A day 56 / HAMA Day 1. Thus, larger numbers equal a greater reduction in anxiety.
Time Frame: % change in anxiety from Day 1 to Day 56 (week 8)
Population: Only participants completing the protocol are included in the analysis. Only participants in the Depressed group were analyzed for change in anxiety symptoms.
Measure: Mean (Standard Deviation); unit: percentage of change in anxiety
Arm/Group | Depressed
Number analyzed (Participants) | 12
percentage of change in anxiety | .3988 (.43)
Statistical Analysis 1: Comparison: Depressed; Test type: Other; p < .006, t-test, 2 sided; Single group t-test

ADVERSE EVENTS:
Arm/Group | Depressed | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/9
Other Adverse Events (participants affected / at risk) | 0/17 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No